CLINICAL TRIAL: NCT06873542
Title: An Open-Label, Dose-Escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Preliminary Efficacy of DC05F01 in Chinese Patients with Advanced or Metastatic Solid Tumors
Brief Title: A Study of DC05F01 in Chinese Patients with Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heronova Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHRC-DC05F01-01
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DC05F01 (Experimental): All enrolled subjects will receive DC05F01 orally. Doses will be escalated from low to high and are coded as Dose Group 1, 2, and 3, with corresponding dosing levels of 1200 mg, 1600 mg, and 2100 mg, respectively.
  Interventions: Drug: DC05F01

INTERVENTIONS:
Drug: DC05F01 — DC05F01 capsule

SUMMARY:
This trial employs a non-randomized, open-label, dose-escalation design to evaluate the safety, tolerability, pharmacokinetic (PK) profile, and preliminary efficacy of DC05F01 in Chinese patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Subjects in each dose cohort will first undergo a single-dose study to assess safety, tolerability, and PK. PK sample collection for the single dose will be conducted over 96 hours. If safety is deemed acceptable after a 5-day observation period (Cycle 0 to Cycle 1 Day 1), subjects will proceed to the multiple-dosing study. The multiple-dosing study will consist of 4-week treatment cycles (daily dosing for 4 weeks, with blood sampling up to 96 hours after the last dose in Cycle 1) (Cycle 1 to Cycle N). The dose limiting toxicity (DLT) observation period will cover the single-dose period and the first cycle of multiple dosing (Cycle 0 + Cycle 1, Day 1 to Day 28). Following this period, subjects will continue with 4-week dosing cycles (Cycle 2 to Cycle N) until they complete six treatment cycles, experience disease progression, develop intolerable toxicity, initiate new anti-tumor therapy, withdraw consent, voluntarily withdraw, die, are lost to follow-up, or encounter other protocol-specified reasons for treatment discontinuation, whichever occurs first. The dose escalation will follow the standard "3+3" design, proceeding from the low-dose group to the high-dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at the time of signing the informed consent form, Chinese male or female.
2. Patients with locally advanced or metastatic solid tumors confirmed by histology and/or cytology, who are refractory to treatment, have failed standard therapy, have no standard treatment options, or for whom standard treatment is not applicable at present.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
4. Presence of at least one measurable or evaluable tumor lesion according to RECIST 1.1 criteria.
5. Expected survival time of ≥3 months.
6. Adequate Organ Function:

   Absolute Neutrophil Count (ANC) >1.5×10^9/L. Hemoglobin (HGB) ≥90 g/L. Platelets (PLT) >100×10^9/L. Total Bilirubin (TBIL) ≤1.5 mg/dL. Albumin (ALB): ≥3 g/dL. Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT)/Alkaline Phosphatase (ALP)/Gamma-Glutamyl Transferase (GGT) ≤2.5 times the upper limit of normal (ULN). If liver metastases are present, AST/ALT/ALP < 5×ULN.

   Serum Creatinine (Scr) ≤1.5×ULN or Creatinine Clearance (CrCl) ≥60 mL/min. Prothrombin Time (PT)/Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN. Serum sodium, potassium, magnesium, calcium, and phosphate levels within normal range or deemed clinically insignificant by the investigator. Supplements to maintain normal electrolyte levels are permitted.
7. Women of childbearing potential must have a negative serum pregnancy test prior to the first dose. Women of childbearing potential are defined as those who have experienced menarche and have not undergone sterilization surgery (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or are not postmenopausal [defined as amenorrhea for at least 12 consecutive months at an appropriate age (e.g., >45 years) with certain clinical manifestations].
8. Men and women of reproductive potential must agree to use reliable contraceptive measures throughout the study period.
9. Ability to understand and voluntarily sign the informed consent form, and willingness to comply with the study's dosing regimen and visit schedule.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, or other anti-tumor treatments within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of the study drug. For nitrosoureas or mitomycin C, this period is extended to 6 weeks.
2. Participated in any other clinical trial and received an investigational drug within 4 weeks before the first dose of the study drug.
3. Adverse effects related to prior chemotherapy, radiotherapy, biological agents, hormonal therapy, or previous investigational treatments have not resolved to ≤Grade 1 (except for alopecia or neurotoxicity of Grade 1-2).
4. Presence of untreated brain metastases or treated brain metastases that have not achieved radiological and clinical stability (i.e., requiring steroid treatment) within 4 weeks before enrollment.
5. Baseline QT/QTc interval prolongation deemed clinically significant by the investigator (calculated using Fridericia's formula, QTc interval >470 ms for females, >450 ms for males).
6. Baseline electrocardiogram (ECG) showing conduction abnormalities or active ischemia deemed clinically significant by the investigator.
7. Presence of uncontrolled or unstable comorbid conditions before enrollment, including but not limited to persistent or active infections, symptomatic congestive heart failure, hypertension, unstable angina, arrhythmias, autoimmune or inflammatory diseases, psychiatric/social disorders, and other conditions that may affect trial compliance as judged by the investigator.
8. Clinically significant gastrointestinal bleeding, bowel obstruction, or gastrointestinal perforation within 6 months before enrollment.
9. Previous allogeneic hematopoietic stem cell or bone marrow transplantation, or previous solid organ transplantation, or current use of immunosuppressive drugs or anti-rejection medications.
10. Need for concomitant use of strong inhibitors or inducers of Cytochrome P450 (CYP) 3A4, CYP1A2, and/or CYP2D6 during the trial.
11. Positive test results for hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody, or anti-treponema pallidum-specific antibody.
12. Pregnant or breastfeeding women.
13. Subjects (or their partners) who plan to conceive during the trial or within 3 months after the last dose of the study drug.
14. Subjects deemed unsuitable for the trial by the investigator due to other reasons (such as abnormal laboratory test results, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 6 months
  Incidence and severity of adverse events as assessed by CTCAE Version 5.0

SECONDARY OUTCOMES:
PK profile of DC05F01 | From time zero up to 96 hours post-dose
  Peak Concentration (Cmax): The maximum plasma concentration of the drug.
PK profile of DC05F01 | From time zero up to 96 hours post-dose
  Area Under the Curve from Time Zero to the Last Measurable Concentration (AUC0-t): The area under the plasma concentration-time curve from time zero to the last measurable concentration.
PK profile of DC05F01 | From time zero up to 96 hours post-dose
  Area Under the Curve from Time Zero Extrapolated to Infinity (AUC0-∞): The area under the plasma concentration-time curve from time zero extrapolated to infinity.
PK profile of DC05F01 | From time zero up to 96 hours post-dose
  Time to Reach Peak Concentration (Tmax): The time at which the peak plasma concentration is reached.
PK profile of DC05F01 | From time zero up to 96 hours post-dose
  Elimination Half-Life (T1/2): The time required for the plasma concentration to decrease by half.
Overall response rate (ORR) | Up to 6 months
  Overall response rate (ORR) based on RECIST v1.1 as assessed by the investigator
Progression-free Survival (PFS) | Up to 6 months
  Progression-free survival (PFS) based on RECIST v1.1 as assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No